CLINICAL TRIAL: NCT00875511
Title: Effects of a Computer Game on Activity Choices
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Sarah-Jeanne Salvy, Ph.D., University at Buffalo
Other Study IDs: Study #3480
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-04

CONDITIONS: Overweight
Keywords: peer rejection; obesity; amount of food chosen; amount of social time chosen
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The study seeks to discover whether peer rejection increases the value of food relative to peer interaction in overweight individuals. After playing a computer game that randomly simulates peer rejection or peer acceptance, participants will play another computer game that will assess the value of food and social interactions.

Overweight individuals may be more likely to resort to food in moments of distress and less likely to choose to interact with a peer to reestablish their sense of belongingness.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-50
* Adults with a BMI greater than or equal to 18.5
* Adults must report at least a moderate liking of study foods used

Exclusion Criteria:

* Adults should have no psychopathology
* Adults should have no developmental disabilities
* Adults should have no cold or upper respiratory distress that could influence their activities
* Adults should have not be taking medications that could affect their food intake
* Adults should have no dietary restrictions
* Adults should have no food allergies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults between the ages of 18-50
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
amount of food chosen amount of social time chosen

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Salvy, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Division of Behavioral Medicine, Buffalo, New York, United States